CLINICAL TRIAL: NCT04687956
Title: Effect of Lymphatic Microsurgical Preventing Healing Approach (LYMPHA) for Primary Surgical Prevention of Breast Cancer-related Lymphedema
Brief Title: Primary Surgical Prevention of Breast Cancer-related Lymphedema
Acronym: LYMPHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Jeong, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3-2020-0343
Record Dates: First submitted 2020-11-29; First posted 2020-12-29 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Lymphedema; Mastectomy; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LYMPHA (Experimental): LYMPHA procedure is performed in which the lymphatic vessels drained from the arm and the axillary vein are micro-bonded to the side branches.
  Interventions: Procedure: LYMPHA
- Control (Active Comparator): No LYMPHA procedure is performed
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: LYMPHA — Axillary reverse mapping is performed before surgery, axillary lymph node resection is performed, and 'LYMPHA' (Lymphatic microsurgical preventing healing approach) is performed, and the surgery is terminated. Subsequently, the occurrence of lymphedema is followed up.
  Arms: LYMPHA
Procedure: control — In the control group, axillary lymph node resection is performed and the surgery is terminated without additional procedures. Subsequently, the occurrence of lymphedema is followed up.
  Arms: Control

SUMMARY:
Lymphedema refers to edema caused by insufficient drainage of interstitial fluid through the lymphatic circulation system. It occurs mainly in the upper and lower extremities and causes chronic inflammation, and finally fibrous adipose tissue is replaced. In this study, the'LYMPHA' (Lymphatic microsurgical preventing healing approach) procedure, which connects lymphatic vessels drained from the arm to the side branches of the axillary vein, contributes to the prevention of lymphedema in patients undergoing axillary lymph node dissection for breast cancer. Investigator aim to help patients' quality of life by prospectively analyzing the effects and applying them to clinical practice, reducing the incidence of lymphedema.

DETAILED DESCRIPTION:
Patients in the LYMPHA group undergo Axillary reverse mapping before the start of surgery, and after axillary lymph node resection, LYMPHA procedure is performed in which the lymphatic vessels drained from the arm and the axillary vein are micro-bonded to the side branches.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 19 years old
2. Patients who are expected to undergo surgery under the diagnosis of breast cancer, and are determined to undergo axillary lymph node dissection before surgery.

Exclusion Criteria:

1. Patients with vascular and lymph-related diseases
2. Patients with a history of surgical treatment or trauma to both arms and axillary
3. Patients with a history of receiving radiation treatment in both arms, chest, and axilla
4. Patients with confirmed systemic metastasis with stage 4 breast cancer
5. Pregnant and lactating patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patient
Enrollment: 72 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of lymphedema | 2 years after surgery
  To compare the incidence of lymphedema assessed by UEL index and lymphoscintigraphy at 2 years after the surgery.

SECONDARY OUTCOMES:
UEL index | 2 years after surgery
  To compare the UEL index
Changes in Lymphoscintigraphy | 2 years after surgery
  To compare the changes in lymphoscintigraphy presented by the change of transport index (TI)
Incidence of lymphedema | 5 years after surgery
  To compare the incidence of lymphedema assessed by UEL index and lymphoscintigraphy at 5 years after the surgery.
5-year recurrence rate | 5 years after surgery
  To compare the recurrence rate
5-year overall survival rate | 5 years after surgery
  To compare the overall survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea